CLINICAL TRIAL: NCT07233525
Title: Culturally Adapted Home-Based Intervention to Improve Language and Cognitive Development in Arab Toddlers in Israel: A Randomised Controlled Trial
Brief Title: Home-Based Language and Cognitive Intervention for Arab Toddlers in Israel
Acronym: CAHBI-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0159-22-HYMC
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Enhancing Early Language and Cognitive Development in Toddlers Through a Culturally Adapted Home-based Parent Intervention
Keywords: Early childhood intervention; Home-based intervention; Language development; Cognitive development; Developmental delay; Parents responsiveness; Low SES intervention; ecological; CAT-CLAMS; Communicative Development Inventories (CDI); Arabic
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors conducting post-intervention evaluations will be blinded to group allocation. Participants and interventionists cannot be blinded due to the nature of the home-based behavioural intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child language and cognitive development (Experimental): Eight weekly home-based sessions focusing on:
  1. Optimising the physical environment
  2. Following the child's interests in play
  3. Enhancing parental responsiveness during exploration, play, and communication
  4. Integration into daily routines and story time
  Interventions: Behavioral: Culturally Adapted Parent-Implemented Intervention
- Child Health Education (Active Comparator): Eight weekly sessions on topics such as healthy sleep, nutrition, toilet training, vaccinations, and safe routines. Same schedule and duration as the intervention arm but without language or cognitive stimulation.
  Interventions: Behavioral: Child Health Education Sessions

INTERVENTIONS:
Behavioral: Culturally Adapted Parent-Implemented Intervention — A culturally adapted, parent-implemented home program designed to enhance toddlers' language, communication, and problem-solving skills. Trained facilitators deliver eight weekly 30-45-minute sessions in the family's home. Sessions focus on three everyday contexts-play, daily routines, and shared story time. Parents are guided to optimise the home environment, follow the child's interests, and use responsive interaction strategies such as joint attention, labelling, expansions, imitation, questioning, and scaffolding. Sessions progress from play-based interaction to integration into routines and storytelling.
  Arms: Child language and cognitive development
Behavioral: Child Health Education Sessions — Eight weekly home-based sessions delivered by trained facilitators, focusing on child health and wellbeing (nutrition, sleep, safety, vaccination, and toilet training). Sessions match the intervention arm in frequency, duration, and contact time but do not include language or cognitive stimulation components.
  Arms: Child Health Education

SUMMARY:
This study evaluates the effectiveness of a culturally adapted, home-based program designed to improve language and cognitive development in Arab toddlers in Israel. Families with children aged 18-36 months will participate in eight weekly sessions delivered in their homes. The intervention teaches parents strategies to enhance their child's language, communication, and problem-solving through play, daily routines, and story time. A comparison group will receive eight sessions on child health promotion (nutrition, sleep, safety, etc.). Child outcomes will be assessed using the Clinical Adaptive Test/Clinical Linguistic and Auditory Milestone Scale (CAT-CLAMS) and the Arabic Communicative Development Inventories (CDI). This research aims to provide an evidence-based, scalable model for early childhood interventions in disadvantaged populations.

DETAILED DESCRIPTION:
Arab children aged 0-3 years in Israel are considered at high risk for cognitive, linguistic, and educational disadvantages due to structural and socio-cultural factors, including poverty, geographic and social marginalisation, and underutilization of daycare and health services. Despite evidence that early intervention supports language and cognitive development, few culturally adapted, evidence-based programs have been evaluated in this population.

This study evaluates a home-based, culturally adapted early childhood intervention designed to enhance language, communication, and problem-solving skills in Arab toddlers (18-36 months). The intervention is guided by Bronfenbrenner's ecological framework and emphasises caregiver responsiveness, considering the child's developmental characteristics, the caregiver's behaviour, and the family's physical and social environment.

The program consists of eight weekly sessions delivered in the family's home, focusing on three contexts: play, daily routines, and shared story time. Parents are guided to optimise the home environment, follow the child's interests, and use responsive behaviours such as joint attention, labelling, expansions, imitation, questioning, and scaffolding. Sessions progress from play-based strategies to generalisation in routines and storybook reading.

Families randomised to the control arm receive eight home-based health-promotion sessions, matched in frequency and duration, covering topics such as nutrition, sleep routines, vaccinations, and toilet training. This serves as an attention-control condition without direct cognitive or language stimulation.

Participants include children aged 18-36 months with no severe medical conditions, birth weight ≥1500g, and scores at the lower end of the normative range on the CAT-CLAMS (approximately -1 to -2 SD below the mean). Caregivers must agree to participate and must not show moderate-to-severe depressive symptoms (PHQ-9 ≥10). Recruitment will occur via community healthcare centres ("well-baby" clinics).

Primary outcomes are changes in language and cognitive development, assessed with the CAT-CLAMS and the Arabic adaptation of the MacArthur-Bates Communicative Development Inventories (CDI). Secondary outcomes include caregiver-reported developmental concerns measured by the Parents' Evaluation of Developmental Status (PEDS). Assessments occur at baseline and one month post-intervention by blinded evaluators.

This trial will provide critical evidence regarding culturally adapted, parent-implemented interventions in marginalised populations. By addressing the ecological context of Arab families in Israel, the program aims to strengthen early language and cognitive skills, reduce risk of later academic and social difficulties, and contribute to the evidence base for scalable early developmental interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-36 months
* Birth weight ≥1500 g
* No significant sensory impairments or severe medical conditions
* CAT-CLAMS scores at the lower end of the normative range (approximately -1 to 1.5 SD below mean)
* Caregiver willing to participate in eight home sessions
* Caregiver without moderate or severe depressive symptoms (PHQ-9 < 10)

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Arabic-CDI total vocabulary score | Baseline to 1-month post-intervention
  Parent-reported receptive and expressive vocabulary.
Change in the CAT-CLAMS total score | Baseline to 1-month post-intervention
  : Measures language, communication, problem-solving, and adaptive behaviours.

SECONDARY OUTCOMES:
Change in PEDS parental concern score | Baseline to 1-month post-intervention
  Parent reported developmental concerns

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Centres - Northern, Central, and Southern Israel, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slobodin O, et al. (2021). Cultural adaptation of early childhood interventions: A systematic review. Early Childhood Research Quarterly, 57, 1-14.
- Available data/document: Study Protocol — https://osf.io/ryq6k/overview?view_only=82691366adfe4dd3999bfba95ce6466d — The full study protocol